CLINICAL TRIAL: NCT00070161
Title: Donepezil and EGb761 in Improving Neurocognitive Function in Patients Who Have Previously Undergone Radiation Therapy for Primary Brain Tumor or Brain Metastases
Brief Title: Phase II Studies Of Donepezil And Ginkgo Biloba In Irradiated Brain Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: REBACCCWFU-97100; U10CA081851 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Radiation Toxicity
Keywords: radiation toxicity; adult mixed glioma; adult central nervous system germ cell tumor; adult brain stem glioma; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult choroid plexus tumor; adult tumors metastatic to brain; adult anaplastic oligodendroglioma; adult anaplastic astrocytoma; adult pilocytic astrocytoma; adult subependymoma; adult meningeal hemangiopericytoma; adult ependymoblastoma; adult anaplastic ependymoma; adult pineoblastoma; adult pineocytoma; adult myxopapillary ependymoma; adult glioblastoma; adult grade III meningioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Radiation Injuries; Glioma; Craniopharyngioma; Medulloblastoma; Meningioma; Choroid Plexus Neoplasms; Brain Neoplasms; Oligodendroglioma; Astrocytoma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Ependymoma; Pinealoma; Glioblastoma; Gliosarcoma | interventions — Ginkgo biloba extract; Donepezil; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: EGb761
Drug: donepezil hydrochloride
Procedure: cognitive assessment

SUMMARY:
RATIONALE: Donepezil and EGb761 may be effective in improving neurocognitive function (such as thinking, attention, concentration, and memory) and may improve quality of life in patients who have undergone radiation therapy to the brain.

PURPOSE: This phase II trial is studying how well donepezil or EGb761 works in improving neurocognitive function in patients who have undergone radiation therapy for primary brain tumor or brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of donepezil or EGb761 on neurocognitive function in patients who underwent radiotherapy for a primary brain tumor or brain metastases at least 6 months before study registration.

Secondary

* Determine the toxicity of these drugs in these patients.
* Determine the quality of life of patients treated with these drugs.
* Quantify the extent of radiation-induced white matter disease and temporal lobe atrophy in patients treated with these drugs.

OUTLINE: This is an open-label, multicenter study.

* Group 1 (closed to accrual 10/09/03): Patients receive oral donepezil once daily for 24 weeks.
* Group 2: Patients receive oral EGb761 three times daily for 24 weeks. In both groups (group 1 closed to accrual 10/09/03), treatment continues in the absence of unacceptable toxicity.

In both groups (group 1 closed to accrual 10/09/03), quality of life and neurocognitive assessment is performed at baseline and at weeks 6 (group 1 only), 12, 24, and 30.

Patients are followed at 6 weeks.

PROJECTED ACCRUAL: A total of 70 patients (35 per treatment group) will be accrued for this study within 9.5 months. (Group 1 closed to accrual 10/09/03)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary brain tumor or brain metastases, meeting 1 of the following criteria:

  * No radiographic evidence of disease
  * Stable disease, defined as no tumor progression within the past 3 months
* Previously treated with 1 course of localized or whole brain radiotherapy of at least 3,000 cGy at least 6 months before study registration

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 30 weeks

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* Concurrent steroid therapy allowed if on stable or decreasing dose

Radiotherapy

* See Disease Characteristics
* No concurrent cranial radiotherapy

Surgery

* No concurrent surgery

Other

* More than 3 months since prior donepezil or EGb761
* No concurrent donepezil (group 2 only)
* No concurrent EGb761 (group 1 only) (closed to accrual 10/09/03)
* No concurrent anticoagulants (e.g., aspirin, dipyridamole, heparin, warfarin, or enoxaparin) (group 2 only)
* No concurrent monoamine oxidase inhibitors (e.g., phenelzine or tranylcypromine)
* No other concurrent therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2001-07-01 (Actual); Primary Completion 2005-05-01 (Actual); Study Completion 2012-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaw EG, Rosdhal R, D'Agostino RB Jr, Lovato J, Naughton MJ, Robbins ME, Rapp SR. Phase II study of donepezil in irradiated brain tumor patients: effect on cognitive function, mood, and quality of life. J Clin Oncol. 2006 Mar 20;24(9):1415-20. doi: 10.1200/JCO.2005.03.3001. PMID 16549835